CLINICAL TRIAL: NCT00621634
Title: Randomized, Double-Blind, Placebo-Controlled Trial on the Efficacy of Omega-3 Supplementation With Docosahexaenoic Acid (DHA) on Tardive Dyskinesia
Brief Title: Efficacy of Docosahexaenoic Acid on Tardive Dyskinesia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Université de Montréal (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other)
Responsible Party: Pierre Blanchet/principal investigator, University of Montreal Hospital Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HD06.067
Record Dates: First submitted 2008-02-12; First posted 2008-02-22 (Estimated); Last update posted 2008-02-22 (Estimated); Status verified 2007-09

CONDITIONS: Tardive Dyskinesia
Keywords: Tardive dyskinesia; Schizophrenia; Essential fatty acids
MeSH Terms: conditions — Tardive Dyskinesia; Schizophrenia | interventions — Fish Oils

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Active treatment with omega-3 fish oil capsules (1 g each capsule, 50% DHA), 6 capsules each day for 12 weeks
  Interventions: Dietary Supplement: Omega-3 fish oil capsules (including DHA)
- 2 (Placebo Comparator): Matching placebo treatment
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Omega-3 fish oil capsules (including DHA) — Fish oil capsules of 1000 mg ea., including DHA 460-540 mg/capsule 2 capsules TID daily at mealtime for 12 consecutive weeks
  Other Names: 0355EEPB1000CT (Ocean Nutrition Canada)
  Arms: 1
Dietary Supplement: Placebo — Corn/Soybean (1:1) placebo 1000 mg capsules 2 capsules TID daily at mealtime for 12 consecutive weeks
  Other Names: Placebo1000 (Ocean Nutrition Canada)
  Arms: 2

SUMMARY:
Tardive dyskinesia (TD) is a well-known complication of antipsychotic drug therapy in individuals treated for mental disorders such as schizophrenia. It typically consists of purposeless, involuntary movements involving the mouth area or the trunk and limb muscles, occurring within months or years of drug use. The annual incidence of TD in the population treated with antipsychotic drugs is between 1-5%, but the risk is 5-fold greater in older individuals. Once triggered, TD is often irreversible and untreatable. Its cause is unknown, but an imbalance between chaotic mechanisms triggered by the drugs and natural protective factors fighting against these may provide an explanation. One way to activate this protective response is to supplement the diet with high doses of essential fatty acids of the omega-3 class, which constitute a critical component of nerve cell membranes. Using this strategy, one research team showed a 50% reduction in the severity of TD-like movements in mice treated with docosahexaenoic acid (DHA). We hypothesize that DHA supplements can do the same in patients living with schizophrenia displaying TD movements. Forty (40) subjects between 30-75 years of age will be recruited. The participants will be randomized and equally distributed in two groups to take either DHA capsules (3 grams a day) or matching placebo for 12 weeks, after providing informed consent, and TD will be measured with a magnetic tracker system and clinical scales. The finding of a beneficial effect with DHA against TD would improve the quality of life for thousands of patients under long-term antipsychotic drug treatment.

DETAILED DESCRIPTION:
Background

Tardive dyskinesia (TD) is a well-known complication of antipsychotic drug (APD) therapy in individuals treated for mental disorders such as schizophrenia. It typically consists of purposeless, involuntary movements involving the oro-facial area, trunk, and/or limb muscles, occurring within months or years of APD use. Twisting and protruding movements of the tongue, lip smacking and puckering, and chewing movements, are often observed. Oral dyskinesia may cause pain, traumatic lesions, tooth wear, impaired retention of prosthetic devices, chewing difficulty, dysphagia, speech impairment, as well as social embarrassment. The annual incidence of TD in the population treated with these drugs is between 1-5%, but the risk in older individuals is 5-fold greater. The second-generation ("atypical") APDs have substantially reduced the short-term risk of TD, but the annual incidence of TD in older individuals taking these drugs remains comparable to that of younger adults treated with first-generation APDs. The cause of TD is unknown. Since all APDs are blockers of dopamine D2 receptors in the brain, researchers hypothesized that these receptors (or their signaling pathways) become supersensitive in such a way to promote TD. APDs also modulate the expression of a number of brain factors belonging to the nuclear receptor family, including Retinoid X Receptors (RXR) and Nur77, which are overexpressed following chronic APD treatment. These factors, seemingly mounting an adaptive response to fend off adverse drug reactions such as TD, may become incompetent or insufficient over time in those individuals developing TD. One way to activate this response is to supplement the diet with high doses of essential fatty acids of the omega-3 class, which constitute a critical component of nerve cell membranes and modulate a variety of brain receptors. Once triggered, TD is often irreversible and untreatable. However, one team recently showed a 50% reduction in the severity of TD-like movements in mice treated with docosahexaenoic acid (DHA).

Hypothesis

Since there is an apparent close relationship between retinoid receptors and dopamine systems in the human brain and DHA is a RXR agonist, our working hypothesis is that DHA will reduce TD intensity in patients living with schizophrenia by increasing the transcriptional activity along these pathways.

Objective

To evaluate the clinical impact of DHA on the intensity of TD in humans.

Study design

Forty (40) subjects between 30-75 years of age will be recruited. The participants will be randomized and equally distributed in parallel groups to take either DHA (3 grams a day) or matching placebo capsules for 12 weeks, after providing informed consent. The study will use questionnaires, venous blood sampling, as well as clinical scales, to monitor the psychiatric condition, the lipid profile, and TD intensity at the beginning and end of the study. Brief and simple tasks will also be completed with a motion analysis system using magnetic sensors in order to measure body movements and TD with accuracy.

Outcome

The finding of a beneficial effect with DHA against TD would improve the quality of life for thousands of patients under long-term APD treatment.

ELIGIBILITY:
Inclusion Criteria:

* chronic schizophrenia patients under long-term antipsychotic drug treatment, stable for at least 3 months before study entry;
* presence of tardive dyskinesia following Schooler-Kane research criteria (mild intensity (2/4 points) in at least two body segments, or moderate intensity (3∕4 points) for at least one body segment);
* patients capable to understand the goals and procedures of the study, and to provide informed consent;
* women of childbearing age will be requested to use an effective contraceptive method throughout the study.

Exclusion Criteria:

* subjects with medical conditions susceptible to significantly increase the risk of adverse effects, or to interfere with the conduct of the study; in particular, those with a history of coronary artery disease, pancreatitis, diabetes, coagulation disorders, or hemorrhagic conditions;
* those regularly taking aspirin, anticoagulants, or oral lipid-lowering agents;
* those with fasting baseline triglyceride values >4.0 mmol/L, or with cholesterol values >8 mmol/L ;
* those intolerant or allergic to fish, seafood, or any other substance contained in the study medication or matching placebo;
* those who have abused illegal street drugs during the past year;
* those unlikely to comply with the study requirements;
* those who consume natural health products of marine or vegetable source, containing omega-3 essential fatty acids;
* women who are pregnant or breastfeeding.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-02; Primary Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Clinical rating scales (AIMS, St.Hans) | Baseline, Week 2, Week 14

SECONDARY OUTCOMES:
Quantitative motor testing (kinematic parameters) | Baseline, Week 14
Monitoring of psychopathology (Neuro-Psychiatric Inventory, Positive and Negative Syndrome Scale, Calgary Depression Scale for Schizophrenia) | Baseline, Week 2, Week 14
Erythrocyte membrane phospholipid profile (gas chromatography) | Baseline, Week 14

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Louis-H.-Lafontaine Hospital, Montreal, Quebec
  - Notre-Dame Hospital/CHU Montreal, Montreal, Quebec

REFERENCES:
- [Background] Ethier I, Kagechika H, Shudo K, Rouillard C, Levesque D. Docosahexaenoic acid reduces haloperidol-induced dyskinesias in mice: involvement of Nur77 and retinoid receptors. Biol Psychiatry. 2004 Oct 1;56(7):522-6. doi: 10.1016/j.biopsych.2004.06.036. PMID 15450789
- [Background] Beaudry G, Langlois MC, Weppe I, Rouillard C, Levesque D. Contrasting patterns and cellular specificity of transcriptional regulation of the nuclear receptor nerve growth factor-inducible B by haloperidol and clozapine in the rat forebrain. J Neurochem. 2000 Oct;75(4):1694-702. doi: 10.1046/j.1471-4159.2000.0751694.x. PMID 10987852
- [Background] Langlois MC, Beaudry G, Zekki H, Rouillard C, Levesque D. Impact of antipsychotic drug administration on the expression of nuclear receptors in the neocortex and striatum of the rat brain. Neuroscience. 2001;106(1):117-28. doi: 10.1016/s0306-4522(01)00248-2. PMID 11564422